CLINICAL TRIAL: NCT04994613
Title: Use of an Adaptive Sensory Environment in Autism Spectrum Disorder (ASD) Patients in the Perioperative Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dayton Children's Hospital (Other)
Collaborators: The Robert C. Cohn Research Endowment (Unknown)
Responsible Party: Principal Investigator, Sean Antosh, Pediatric Anesthesiologist, Dayton Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 21-037
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder; Anesthesia; Procedural Anxiety; Sensory Processing Disorder
Keywords: Pediatric Anesthesia; Autism Spectrum Disorder; Procedural Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The control group will be standard practice with no sensory adaptive environment and the intervention group with be a sensory adaptive environment. Patients will be randomized in varying block sizes using a random number generator to ensure equal numbers in each group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The random allocation, block sizes, and block sequences will be concealed from study personnel and each patient until the time a patient is assigned to a group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The patient will be reserved a standard room in the preoperative area of main campus. This room will not include any additional sensory equipment. The child will be allowed to use any comfort items the family brought with them or offered a hospital iPad, as is current practice for all outpatient surgery patients.
- Sensory Adaptive Environment Group (Experimental): One of the three dedicated adaptive sensory rooms in the preoperative area of main campus will be set up by nursing and child life staff in accordance with the patient's coping plan and individual needs regarding sound, light, activity level, and other stimuli. The equipment may include a portable popcorn tube with fiberoptic cart, handheld marble panel, color changing floor tiles, other sensory friendly objects, and individual sensory toys. This room will be set up prior to the patient's arrival the day of surgery and reserved for their use.
  Interventions: Other: Sensory adaptive environment

INTERVENTIONS:
Other: Sensory adaptive environment — A dedicated, private room that is set up in accordance with the patient's coping plan and individual needs regarding sound, light, activity level, and other stimuli.
  Arms: Sensory Adaptive Environment Group

SUMMARY:
The objective of this study is to prospectively examine the preoperative anxiety scores of ASD patients in an adaptive sensory environment. Additionally, the investigators aim to determine the relationship of severity of sensory integration in ASD patients and their preoperative anxiety scores. The study will also study the family satisfaction with tailored care of their ASD child in the peri-operative environment.

DETAILED DESCRIPTION:
At Dayton Children's, all patients with autism or other developmental delays are called prior to the day of surgery by child life specialists to obtain a coping plan to be entered into the EHR. Those patients that meet the criteria will be approached via telephone call 24-48 hours prior to procedure by the research team to describe the study and gauge interest in participating.

The pilot study will recruit a total of sixty patients in two parallel groups randomized to 1:1 allocation: control group (standard practice with no sensory adaptive environment) or intervention group (sensory adaptive environment). Patients will be randomized in varying block sizes using a random number generator to ensure equal numbers in each group. The random allocation, block sizes, and block sequences will be concealed from study personnel and each patient until the time a patient is assigned to a group.

In the preoperative area of main campus perioperative services there are three dedicated adaptive sensory friendly rooms for patients to await surgery. For the sensory adaptive environment, the room will be set up in accordance with the patient's coping plan and individual needs regarding sound, light, activity level, and other stimuli. The equipment may include a portable popcorn tube with fiberoptic cart, handheld marble panel, color changing floor tiles, other sensory friendly objects, and individual sensory toys.

After registration and informed consent, the patient will be placed in either a standard preoperative room (control) or the dedicated sensory rooms (intervention) in the preoperative surgery area based on prior randomization. The patient's behaviors will be recorded by a research assistant at three time points (registration, nursing intake in preoperative room, and immediately prior to transition to operating room) by utilizing the validated modified Yale Preoperative Anxiety Scale (mYPAS). The mYPAS is the most widely used tool for assessing preoperative anxiety in children. The total score on the mYPAS will be the primary outcome for the study.

In addition to the mYPAS measurements, the patient will be evaluated in the operating room utilizing the validated Child Induction Behavioral Assessment Scale (CIBA). The CIBA is a 3-category behavioral assessment for documenting children's behavioral responses to induction of anesthesia. The 3 categories, Smooth, Moderate, and Difficult have associated behavioral descriptions that are scored at the time of anesthesia induction. The CIBA will be evaluated by the assigned anesthesia staff and documented in the EHR, as current standard practice.

While the patient is in the procedure, families will fill out two questionnaires in the waiting room. The first is a 23-item questionnaire (Patient Experience Study Survey) regarding the patient preoperative experience.

The second questionnaire is the Short Sensory Profile 2 (SSP-2), which assesses the patient's sensory processing abilities. The SSP-2 score will be used as a surrogate for the severity of sensory sensitivity in the study patient.

In addition to the SSP-2, the following independent variables will be extracted from the medical record: patient demographics (sex, age, weight), ASA score designated by anesthesiologist, diagnosis and health history, procedure, home medications, preoperative medications including dose and route, intraoperative medications, event times and durations (including preoperative wait time, transport to OR time, induction to anesthesia ready, case length, & recovery time), and first recovery room pain score (documented by PACU RN via FLACC score).

ELIGIBILITY:
Inclusion Criteria:

1. Formal diagnosis of Autism Spectrum Disorder, Asperger's Syndrome, or pervasive developmental disorder NOS
2. Presenting for outpatient surgery at Dayton Children's Hospital main campus

Exclusion Criteria:

1. A coping plan is not able to be obtained prior to day of surgery
2. An American Society of Anesthesiology (ASA) risk score greater than 3
3. Non-English speaking
4. Refusal of participation by guardian

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Examine the preoperative anxiety scores of ASD patients in an adaptive sensory environment. | From procedural registration to induction of anesthesia (approximately 1-2 hours)
  The validated modified Yale Preoperative Anxiety Scale (mYPAS) will be utilized to assess anxiety and behaviors at three time points in the preoperative process, to include registration in the surgery lobby, preoperative nurse intake in the individual room, and immediately prior to transition to operating room.mYPAS consists of 5 items; 4 of the items (Activity, Emotional Expressivity, State of Apparent Arousal, and Use of Parent) are rated on scales of 1-4, and 1 item (Vocalizations) is rated on a scale of 1-6. The total score is determined by dividing each item rating by its highest possible rating, summing the results, dividing by 5, and then multiplying by 100. Total scores can range from 23.33 to 100, with higher scores representing greater anxiety.

SECONDARY OUTCOMES:
Determine the relationship of severity of sensory integration in ASD patients and their preoperative anxiety scores. | Obtained during patient's procedure.
  Patient's primary caregiver will complete the Short Sensory Profile 2 (SSP-2), which assesses the patient's sensory processing abilities. The SSP-2 score will be used as a surrogate for the severity of sensory sensitivity in the study patient. The SSP-2 consists of 34 behavioral items measured on 5-point Likert scales from 1 = almost never to 5 = almost always. Items are divided into 4 quadrants for scoring, Seeking (7 items), Avoiding (9 items), Sensitivity (10 items), and Registration (8 items) based on Dunn's Sensory Processing Framework. Two subscale scores, Sensory Processing and Behavioral Responses Associated with Sensory Processing, as well as total scores are also determined. Raw scores are compared to a normal curve and Sensory Profile 2 Classification System developed from a normative sample.
Explore family satisfaction with tailored care of their ASD child in the peri-operative environment. | Obtained during patient's procedure.
  Patient's primary caregiver will document on a 23-item questionnaire (Patient Experience Study Survey) regarding the patient preoperative experience. The first section includes yes/no questions regarding parent's discussions with Dayton Children's Child Life prior to the day of surgery in developing the coping plan. The second and third sections use positively worded statements measured on 5-point Likert scales from 1 = strongly disagree to 5 = strongly agree. These two sections discuss the preoperative holding room and environment on the day of surgery (9 items), and how the perioperative team related to the patient (5 items). Total scores across all items will be determined, as well as scores within each of the 3 sections. A final item will ask the family to rate the overall experience on a 10-point scale from 1 = very dissatisfied to 10 = very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Antosh, MD, Principal Investigator — Dayton Children's Hospital
Locations (1):
- Dayton Children's Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott AB, Holley AL, Ross AC, Soleta AO, Koh JL. A prospective study comparing perioperative anxiety and posthospital behavior in children with autism spectrum disorder vs typically developing children undergoing outpatient surgery. Paediatr Anaesth. 2018 Feb;28(2):142-148. doi: 10.1111/pan.13298. Epub 2017 Dec 10. PMID 29226493
- [Background] Arnold B, Elliott A, Laohamroonvorapongse D, Hanna J, Norvell D, Koh J. Autistic children and anesthesia: is their perioperative experience different? Paediatr Anaesth. 2015 Nov;25(11):1103-10. doi: 10.1111/pan.12739. Epub 2015 Sep 4. PMID 26338278
- [Background] Taghizadeh N, Davidson A, Williams K, Story D. Autism spectrum disorder (ASD) and its perioperative management. Paediatr Anaesth. 2015 Nov;25(11):1076-84. doi: 10.1111/pan.12732. Epub 2015 Aug 6. PMID 26248302
- [Background] Swartz JS, Amos KE, Brindas M, Girling LG, Ruth Graham M. Benefits of an individualized perioperative plan for children with autism spectrum disorder. Paediatr Anaesth. 2017 Aug;27(8):856-862. doi: 10.1111/pan.13189. Epub 2017 Jun 15. PMID 28618130
- [Background] Cermak SA, Stein Duker LI, Williams ME, Dawson ME, Lane CJ, Polido JC. Sensory Adapted Dental Environments to Enhance Oral Care for Children with Autism Spectrum Disorders: A Randomized Controlled Pilot Study. J Autism Dev Disord. 2015 Sep;45(9):2876-88. doi: 10.1007/s10803-015-2450-5. PMID 25931290
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Winterberg AV, Ding L, Hill LM, Stubbeman BL, Varughese AM. Validation of a Simple Tool for Electronic Documentation of Behavioral Responses to Anesthesia Induction. Anesth Analg. 2020 Feb;130(2):472-479. doi: 10.1213/ANE.0000000000003945. PMID 30531219
- [Background] Simpson K, Adams D, Alston-Knox C, Heussler HS, Keen D. Exploring the Sensory Profiles of Children on the Autism Spectrum Using the Short Sensory Profile-2 (SSP-2). J Autism Dev Disord. 2019 May;49(5):2069-2079. doi: 10.1007/s10803-019-03889-2. PMID 30673910
- [Background] Chojnicka I, Pisula E. Adaptation and psychometric properties of the Polish version of the Short Sensory Profile 2. Medicine (Baltimore). 2019 Nov;98(44):e17689. doi: 10.1097/MD.0000000000017689. PMID 31689792
- [Background] Hanna AH, Ramsingh D, Sullivan-Lewis W, Cano S, Leiter P, Wallace D, Andrews G, Austin B, Applegate RL 2nd. A comparison of midazolam and zolpidem as oral premedication in children, a prospective randomized double-blinded clinical trial. Paediatr Anaesth. 2018 Dec;28(12):1109-1115. doi: 10.1111/pan.13501. Epub 2018 Oct 17. PMID 30328648
- [Background] Kerimoglu B, Neuman A, Paul J, Stefanov DG, Twersky R. Anesthesia induction using video glasses as a distraction tool for the management of preoperative anxiety in children. Anesth Analg. 2013 Dec;117(6):1373-9. doi: 10.1213/ANE.0b013e3182a8c18f. PMID 24257388
- [Background] Lee J, Lee J, Lim H, Son JS, Lee JR, Kim DC, Ko S. Cartoon distraction alleviates anxiety in children during induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1168-73. doi: 10.1213/ANE.0b013e31824fb469. Epub 2012 Sep 25. PMID 23011563
- [Derived] Antosh S, Drennan C, Stolfi A, Lawson R, Huntley E, McCullough-Roach R, Hill M, Adelekan T, Vachhrajani S. Use of an adaptive sensory environment in patients with autism spectrum disorder (ASD) in the perioperative environment: a parallel, randomized controlled trial. Lancet Reg Health Am. 2024 Apr 18;33:100736. doi: 10.1016/j.lana.2024.100736. eCollection 2024 May. PMID 38645550